CLINICAL TRIAL: NCT05023694
Title: Identification And Prevention Of Risk Related Assistance During Stabilization Operations And Resuscitation In Newborns At Birth
Brief Title: Risk Related Assistance During Stabilization In Newborns At Birth
Status: Completed | Type: Observational
Sponsor: Manuel Sanchez Luna (Other)
Responsible Party: Sponsor-Investigator, Manuel Sanchez Luna, Dr., Hospital General Universitario Gregorio Marañon
Organization: Hospital General Universitario Gregorio Marañon (Other)
Other Study IDs: Neo.Segur2
Record Dates: First submitted 2016-04-23; First posted 2021-08-26 (Actual); Last update posted 2021-08-26 (Actual); Status verified 2021-08

CONDITIONS: Infant, Newborn
Keywords: Newborn; adverse events; video record; resuscitation
MeSH Terms: interventions — Videotape Recording

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes

GROUPS / COHORTS (1):
- Newborn reanimated video recordings: Newborns, requiring stabilization at birth in Delivery Room, prior authorization by verbal and written informed consent
  Interventions: Other: Video recordings; Other: Video recordings after corrective measures in adverse events

INTERVENTIONS:
Other: Video recordings — In the first phase it will proceed to completion of the registration system by collecting data revivals and video recordings.
  In a second phase, the video is displayed and analysis of the resuscitation performance will take place. We will identify and make a registration of incidents. At this point the observational descriptive analysis will take place.
  Third phase: to develop preventive measures necessary to limit the number of incidents or to contain or minimize adverse effects resulting thereof: restructure and adapt the protocol.
Other: Video recordings after corrective measures in adverse events — Fourth phase: Training department staff on improvements to optimize performance times protocol using simulation.
  Fifth stage: final implementation of corrective measures of adverse events during the performance resuscitation.
  Sixth stage: successive evaluations of impact of corrective measures. With this evaluation, it will be held another descriptive case series. With the secondary formulate hypothesis after analysis of the errors, the protocol is optimized and measured if errors are minimized: analytical observational prospective cohort study.

SUMMARY:
Approximately 10% of term infants and up to 50% of preterm infants less than 32 weeks require stabilization and / or ventilatory support at the time of transition at birth. Coordination between the rescuer team as well as the precise knowledge of protocol resuscitation maneuvers and indications, the communication of the various professionals involved (gynecologists, pediatricians and anesthesiologists) are critical for proper care and patient stabilization. Common adverse events may hinder or impair the effectiveness of these maneuvers, ventilation, monitoring, ... with consequent worsening in the prognosis of the newborn.

DETAILED DESCRIPTION:
Patient safety is defined as reducing the risk of unnecessary harm associated with healthcare to an acceptable minimum, it is a task for all those involved in the care activity professionals, patients and managers. Since the incidents and adverse events involve a deficit in the quality of care causing damage to users and professionals, and increase healthcare costs, strategies should be to include both the detection and analysis of primary and secondary prevention.

The video recording programs are considered useful to monitor and detect problems during resuscitation and is believed to be useful for improving resuscitation.

HYPOTHESIS Principal: The mismatch in compliance with the guidelines for neonatal resuscitation is the main type of incident during resuscitation due to inadequate stabilization times . The cause of these incidents during resuscitation is varied and not only focuses on personal failure.

As a second hypothesis is that: the implementation of a protocol , after analysis of errors, minimizes by more than 15 % possible incidents and reduces the trip times.

EVALUATION Data collection will be made prospectively. Management during stabilization of the newborn in the delivery room with video is recorded by an independent contributor or fixed camera. Physiological parameters such as air pressure, gas flow , tidal volume , heart rate and oxygen saturation are monitored and recorded in the software monitor respiratory function and analog data FiO2

ELIGIBILITY:
Inclusion Criteria:

* the newborns, who require stabilization at birth in delivery room

Exclusion Criteria:

* reanimation unrecorded with video
* no obtained informed consent

Max Age: 1 Minute | Sex: All | Healthy Volunteers: No
Age Groups: Child
Study Population: The newborns, who require stabilization at birth in delivery room
Sampling Method: Non-Probability Sample
Enrollment: 128 (Actual)
Dates: Start 2016-02; Primary Completion 2016-10 (Actual); Study Completion 2017-02 (Actual)

PRIMARY OUTCOMES:
Identify number and types of adverse events | through study completion, an average of 1 year
  Improve safety and thus the quality of health care in the stabilization and resuscitation of the newborn in Delivery Room by identifying and preventing risks related to patient care.

SECONDARY OUTCOMES:
Preventive measures to limit incidents | through study completion, an average of 1 year
  Optimize a protocol on stabilizing the newborn.
Number of income in Neonatal Unit after resuscitation | through study completion, an average of 1 year
  NICU income
Advanced reanimations | through study completion, an average of 1 year
  Number of advanced resuscitation

CONTACTS AND LOCATIONS:
Overall Officials: Gonzalo Zeballos, Principal Investigator — Gregorio Marañón Hospital
Locations (1):
- HGU Gregorio Marañón Madrid, Madrid, Spain

IPD SHARING:
Plan to Share IPD: No